CLINICAL TRIAL: NCT03829917
Title: Oral Miltefosine Plus Topical Paromomycin In American Cutaneous Leishmaniasis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Fundacion Nacional de Dermatologia (Other)
Collaborators: Hospital Dermatológico de Jorochito (Unknown); Ministerio de Salud de Bolivia, Programa Nacional de Leishmaniasis (Unknown); Alfred Berman Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AB-2018-02
Record Dates: First submitted 2019-01-30; First posted 2019-02-04 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2019-07

CONDITIONS: Cutaneous Leishmaniasis, American
MeSH Terms: conditions — Leishmaniasis, Mucocutaneous | interventions — miltefosine; Paromomycin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Paromomycin and Miltefosine (Experimental): Paromomycin-Aquaphilic cream applied topically once daily for 28 days plus oral miltefosine pills 2.5 mg/day [50 mg tid] for 28 days.
  Interventions: Drug: Miltefosine and Paromomycin
- Miltefosine (Active Comparator): Miltefosine pills alone [2.5 mg/day [50 mg tid] for 28 days. This group will also receive Aquaphilic-vehicle cream for 28 days
  Interventions: Drug: miltefosine
- Paromomycin (Active Comparator): Paromomycin-Aquaphilic cream applied topically once daily for 28 days.
  Interventions: Drug: paromomycin

INTERVENTIONS:
Drug: Miltefosine and Paromomycin — 28 days of miltefosine plus 28 days of Paromomycin cream
  Arms: Paromomycin and Miltefosine
Drug: miltefosine — 28 days of miltefosine
  Arms: Miltefosine
Drug: paromomycin — 28 days of paromomycin creaam
  Arms: Paromomycin

SUMMARY:
Cure rate for L braziliensis bolivian CL has been 70%-80% for standard systemic and local monotherapies. It would benefit patients if cure rates could be consistently >90%, so testing a combination of two treatments is proposed. The most attractive systemic therapy is the only oral agent, miltefosine during 28 days, and the most attractive local therapy is application of Paromomycin cream for 28 days.

DETAILED DESCRIPTION:
Cutaneous leishmaniasis (CL) is endemic in the New World from approximately the US-Mexican border through Central America and the Northern part of South America down to the level of Rio de Janeiro.

L braziliensis CL is perhaps the most important of these diseases, since its natural cure rate is low and it may metastasize, and our group has been evaluating therapies for L braziliensis in Bolivia for some time.

In recent studies at investigator's Bolivian site for the years 2013-2016, the cure rate for L braziliensis CL has been 70%-80% for standard systemic and local therapies. Systemic agents intramuscular pentavalent antimony cured 80% (114 of 143) and oral miltefosine cured 81% (47 of 58). Local injections with pentamidine cured 72% (43 of 60); intralesional antimony cured 70% (21 of 30). In contrast, cryotherapy was ineffective [20% (4 of 20) cured and placebo creams cured 17% (5 of 30) in one report and 10% more recently.

Investigator's have recently evaluated treatment with topical paromomycin cream. Paromomycin-in-Aquaphilic had a cure rate of 77.5% (31 of 40 patients) compared to a cure rate of only 10% (2 of 20 patients) for the Aquaphilic vehicle alone. This remarkably high cure rate, combined with essentially no adverse events (both Paromomycin-Aquaphilic and Aquaphilic vehicle had only grade 1 adverse reactions in 5-10% of patients), makes Paromomycin-Aquaphilic very attractive for Bolivian CL.

It would benefit patients if cure rates could be consistently >90%. Since all the individual therapies, whether systemic, local injections, or local cream, have an approximately 75% cure rate, we propose testing a combination of two treatment. The most attractive systemic therapy is the only oral agent, miltefosine, and the most attractive local therapy is simple application of Paromomycin cream. Thus the present protocol proposes to evaluate the efficacy of miltefosine, 2.5 mg/kg (50 mg tid) for 28 days, plus Paromomycin-Aquaphilic daily for 28 days. The controls will be the two components of this combination used separately: miltefosine alone, Paromomycin-Aquaphilic alone.

ELIGIBILITY:
Inclusion and exlusion Criteria:

* Gender: Male or female
* Age: >12 yrs of age
* Presentation: 1-to-2 ulcerative lesions, each < 30 mm in largest diameter and with a total lesion area <900 mm2.
* Parasitology: Parasitological confirmation of the lesion will be made by visualization or culture of Leishmania from the biopsy or aspirate of the lesion.
* Previous treatment for leishmaniasis:
* No specific or putatively specific therapy (Sb, pentamidine, amphotericin B, miltefosine, imidazoles, allopurinol) in the last 3 months
* Other diseases: No concomitant diseases by history that would be likely in the PI's opinion to interact, either positively or negatively, with treatment.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Size of cutaneous ulcers | 2, 3, 4 and 6 months after the begining of therapy.
  Complete healing of all lesions by 6 months after the beginning of therapy. Thus for a patient to be cured: no lesion could enlarge by 50%, relapse, or heal incompletely; and no new Leishmania-positive lesion can have appeared.

CONTACTS AND LOCATIONS:
Overall Officials: JAIME SOTO, MD, Principal Investigator — Fundación Nacional de Dermatología
Locations (1):
- Hopital, Dermatologico, Jorochito, SC, Bolivia

IPD SHARING:
Plan to Share IPD: No